CLINICAL TRIAL: NCT05233072
Title: Prognostic Impact of Neopterin on Resumption of Walking After a Fracture of the Upper Neck of the Femur in the Elderly
Acronym: MAMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP210718; 2021-A00976-35 (Registry Identifier: DRCB)
Record Dates: First submitted 2021-12-06; First posted 2022-02-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Fracture of Neck of Femur; Resumption of Walking
Keywords: Neopterin
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fracture (Other): Patients with a fracture of the upper neck of the femur
  Interventions: Other: Blood sample
- Control (Other): Patients with no fracture of the upper neck of the femur
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Arm 'Fracture':1 blood sample at D0, D1, D3, D7 and D30 Arm 'Control': 1 blood sample at D0

SUMMARY:
Society faces a major challenge with the management of the health and socio-economic burden caused by acute physical stress in the older population (>75 years). In particular, hip fracture (HF) represents a major health care preoccupation, affecting 1.6 M patients worldwide, resulting in a significant drop of life quality and autonomy. Nowadays, this trauma is still associated with a poor outcome of 20-30% one-year mortality in the elderly. This emphasizes the value of assessing biological factors that may predict clinical outcome after HF. The preliminary work pinpoints a central role of neopterin in loss of autonomy and death. Using HF as an acute stress model that accelerates the progressive course of aging, the aim is to validate neopterin as a predictive biomarker of pernicious clinical outcomes.

DETAILED DESCRIPTION:
Hip fracture (HF) is a common condition affecting an estimated 2 million older people worldwide and that number is increasing by 25% each decade as the population continues to grow. HF has serious clinical consequences due to the associated morbidity, the loss of autonomy in individuals generally autonomous before the event. HF has also been shown to be an independent predictor of a new admission to long-term care, representing an unfavorable outcome with annual costs of four billion in the United States alone. Among the avenues aimed at improving the management of HF, the deployment of perioperative geriatric units (UPOG) has improved the prognosis of patients but their implantations are still unfortunately too marginal. It is therefore in the identification of patients most at risk that research must be focused in order to identify the most vulnerable and target interventions. Today, the decision of admission is made early in the course of care, as soon as their arrival to emergencies, and involves discussion between orthopedist, anesthesiologist and geriatrician. This decision is based on criteria that are still very logistical (place or not), clinical (comorbidities, fragility, severity, etc.) but lacks objective information (no predictive signatures) on resilience post HF.

In this context, prognostic biomarkers would have an important role to play in guiding clinicians. The investigators team has shown that neopterin is a biomarker of inflammation and activation of the immune system secreted during HF and whose increased rate has been associated with mortality at one year post HF as well as with functional recovery on D30 after surgery.

The investigators hypothesize that the neopterin measured at the admission of the elderly patient to the emergency ward for HF could improve the prediction of the resumption of walking without major loss of autonomy at D30 after surgery.

The main objective of the study is to assess whether the plasma neopterin concentration can predict the resumption of walking on D30 after surgery, in elderly patients who have undergone surgery as part of a HF.

ELIGIBILITY:
Inclusion Criteria:

For both arms:

* age over 75
* affiliated to health insurance system
* written informed consent

For arm 'Fracture':

* patient with a fracture of the upper neck of the femur
* hospitalized in emergency in a 'UPOG' unit

For arm 'control':

* hospitalized patient without any acute clinical event

Exclusion Criteria:

For both arms:

* polytrauma
* pathological bone or prothesis fracture
* patient affiliated to 'Aide Médical de l'Etat - AME' insurance
* patient with immunosuppressant treatment (including corticotherapy over 5 mg/d)
* patient with active solid cancer or malignant haemopathy
* patient with auto-immune disease
* refusal to participate in research

For arm 'Fracture':

* patient under justice protection measure except tutorship and guardianship

For arm 'control':

* severe neurocognitive disorders (MMS < 15)
* fracture of the upper neck of the femur in the last year
* patient under justice protection measure

Ages: 75 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Resumption of walking with or without help | Day 30
  Speed walk over 4 meters

SECONDARY OUTCOMES:
Short Physical Performance Battery score | Day 30
  The score is from 0 to 12 based on the result of three exercises: Balance, gait speed and chair stand. 12 means better outcome.
Hand-grip test | Day 30
Measurement of bioimpedancemetry | Day 30
  Measurement of grip strength and of clamp force
Activity of Daily Living score | Day 30
  Score based on a 6-item questionnaire. Each item is rated 0, 0.5 or 1. 1 is the best outcome.
Medical Outcome Study Short Form 12 | Day 30
Number of participants alive | From inclusion to 6 months
Number of participants living at home | Month 6
  Comparison between participants living at home and participants living in an institution

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BODDAERT, MD, Principal Investigator — GH Pitié Salpêtrière - Charles Foix
Locations (1):
- GH Pitié-Salpêtrière / Service de gériatrie, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No